CLINICAL TRIAL: NCT02081508
Title: Consolidation & Interference in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Joshua Sandry, Visiting Scientist Neuropsychology & Neuroscience Research, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R-800-13
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Sclerosis
Keywords: Memory
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Unfilled interference (Experimental): Interference onset: delayed test at 540000 ms
  Interventions: Behavioral: Interference onset
- Early interference (Experimental): Interference onset: delayed test at 0 ms
  Interventions: Behavioral: Interference onset
- Mid interference (Experimental): Interference onset: delayed test at 360000 ms
  Interventions: Behavioral: Interference onset
- Late interference (Experimental): Interference onset: delayed test at 180000 ms
  Interventions: Behavioral: Interference onset

INTERVENTIONS:
Behavioral: Interference onset — Temporal duration of interference onset.

SUMMARY:
The purpose of this research study is to investigate whether minimizing interference improves memory in multiple sclerosis.

DETAILED DESCRIPTION:
The ability to form new long-lasting memories is important for successful independent living and a high quality of life. Roughly half of the individuals diagnosed with Multiple Sclerosis (MS) have difficulty remembering new information and this is likely associated with poor acquisition of new information. There are only a limited number of studies that have investigated memory consolidation in MS. The current study will investigate the role of interference during the consolidation time period of memory formation.

ELIGIBILITY:
Inclusion Criteria:

* If you are between the ages of 18-65.
* If you have a diagnosis of Multiple Sclerosis (MS) or are medically healthy.
* If you have MS, you have not had a flare up of MS symptoms in the past month.
* You do not have other neurological issues such as, Epilepsy or Stroke.
* You do not have a significant history of psychiatric problems or a current diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder .
* You do not have a significant history of drug or alcohol abuse.
* You can read and speak English fluently.
* You are not currently taking steroids.

Exclusion Criteria:

* You are younger than 18 years old.
* You are older than 65 years old.
* You have had a prior stroke or neurological disease other than MS.
* You have a history of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder, Bipolar Disorder.
* You have a significant alcohol or drug abuse history.
* You are currently taking steroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Recall Proportion | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States